CLINICAL TRIAL: NCT04734561
Title: Effects of Respiratory Muscle Training on Quality of Life, Physical and Pulmonary Function and Psychological Status in Patients Who Have Had COVID-19 Disease
Brief Title: Effects of Respiratory Muscle Training in People Who Have Had COVID-19 Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid, Madrid, Spain (Unknown)
Responsible Party: Principal Investigator, Ibai López de Uralde Villanueva, Professor Ibai López de Uralde Villanueva, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20/715-E_BS
Record Dates: First submitted 2020-12-31; First posted 2021-02-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Respiratory Muscle Training; Respiratory Function Test; Quality of Life; Psychosocial Factor
Keywords: COVID-19; Respiratory Muscle Training; Respiratory Function Test; Quality of Life; Psychosocial Factor
MeSH Terms: conditions — COVID-19 | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inspiratory muscle training group (Experimental): Participants will perform an inspiratory muscle training by a threshold device at home, twice a day for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory muscle training group
- Inspiratory muscle training placebo group (Sham Comparator): Participants will perform an inspiratory muscle training by a placebo threshold device at home, twice a day for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory muscle training placebo group
- Inspiratory + expiratory muscle training group (Experimental): Participants will perform an inspiratory and expiratory muscle training by a threshold device at home, twice a day for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory + expiratory muscle training group
- Inspiratory + expiratory muscle training placebo group (Sham Comparator): Participants will perform an inspiratory and expiratory muscle training by a placebo threshold device at home, twice a day for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory + expiratory muscle training placebo group

INTERVENTIONS:
Other: Inspiratory muscle training group — Participants will perform an inspiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Inspiratory muscle training group
Other: Inspiratory muscle training placebo group — Participants will perform an inspiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Inspiratory muscle training placebo group
Other: Inspiratory + expiratory muscle training group — Participants will perform an inspiratory and expiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Inspiratory + expiratory muscle training group
Other: Inspiratory + expiratory muscle training placebo group — Participants will perform an inspiratory and expiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Inspiratory + expiratory muscle training placebo group

SUMMARY:
The main objective of the present study is to observe the short-term effects of respiratory muscle training applied by telerehabilitation on quality of life and exercise tolerance in people who have had the COVID-19 disease. As secondary objectives, the effects on respiratory muscles strength/tolerance, pulmonary function and psychological and cognitive factors.

DETAILED DESCRIPTION:
It is a double-blind randomized clinical trial study. Each participant will be randomly assigned to one of the following groups: 1) Inspiratory muscle training, 2) Placebo Inspiratory muscle training, 3) Inspiratory muscle training + Expiratory muscle training, 4) Placebo Inspiratory muscle training + Expiratory muscle training.

Each exercise training program will be applied twice per day 7 sessions per week during 8 weeks by a threshold device. The evening sessions will be supervised by a physiotherapist through a virtual platform.

Participants received baseline assessments at the beginning of the intervention, at the end of the 4th week, and post-intervention assessments at the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of COVID-19 (SARS-CoV2)
* Hospital admission for COVID-19 in the last 3 months
* Stable phase and home discharge;

Exclusion Criteria:

* Severe cognitive impairment
* Any type of musculoskeletal, neurological, cardiac or respiratory disease where training is contraindicated
* Inability to carry out the training program through telematic supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Change from Baseline Health-related quality of life at 8 weeks
  To evaluate the health-related quality of life of the participants a valid, reliable and generic questionnaire will be used. It consisted of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Exercise tolerance | Change from Baseline Exercise tolerance at 8 weeks
  Exercise tolerance will be evaluated by a test consisted on 30 squats based on three different heart rate measuring moments (resting heart rate, heart rate after exercise, heart rate after longer period) evaluating the speed at which the heart rate increases/decreases.

SECONDARY OUTCOMES:
Maximum respiratory pressures | Change from Baseline Maximum respiratory pressures at 8 weeks
  The maximum respiratory pressures (MIP and MEP) will be measure with a device. This device applies an inspiratory/expiratory load which provides a resistance. The maneuver will be perform in a sitting position. Measuring a minimum of 3 times will be perform, recording the highest value.
Inspiratory muscle endurance | Change from Baseline Inspiratory muscle endurance at 8 weeks
  To measure inspiratory muscle endurance, The subjects inspire from a threshold valve beginning with pressures of 30% of MIP. The threshold pressure is then increased 10% of MIP until the load cannot be tolerated for 2 minutes. The maximum inspiratory mouth pressure that can be tolerated for the full 2-minute interval is considered the peak pressure (Ppeak)
Upper limb muscle strength | Change from Baseline Peripheral muscle strength at 8 weeks
  To measure peripheral muscle strength the isometric strength of the hand and forearm will be evaluated through a valid and reliable tool. Three separate tests will be administered for each arm and the highest value in kilograms will be recorded.
Lung function (forced spirometry) | Change from Baseline Lung function at 8 weeks
  The Spirometry will be perform according to American Thoracic Society criteria and was measured in liters. The maneuver will be perform 3 times and recording the best one.
Cognitive factors | Change from Baseline cognitive factors at 8 weeks
  A validated cognitive scale will be assessed in all study participants with acceptable psychometric properties to evaluate cognitive factors. Unit of Measure: Units on a Scale where higher values represent a greater impact.
Lower limb muscle strength | Change from Baseline Lower limb strength at 8 weeks
  A practical, reliable and valid field test consisted on to complete as many sit-to-stand cycles as possible on a chair during a frame time.
Psychological factors | Change from Baseline Psychological factors at 8 weeks
  A validated anxiety, depression and stress scale will be assessed in all study participants with acceptable psychometric properties to evaluate anxiety and stress factors. Unit of Measure: Units on a Scale where higher values represent a greater impact. These measurements will be aggregated to arrive at one reported value of the impact of Psychological factors.

CONTACTS AND LOCATIONS:
Overall Officials: Ibai López de Uralde Villanueva, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- UComplutenseMadrid, Madrid, Spain

REFERENCES:
- [Background] Disser NP, De Micheli AJ, Schonk MM, Konnaris MA, Piacentini AN, Edon DL, Toresdahl BG, Rodeo SA, Casey EK, Mendias CL. Musculoskeletal Consequences of COVID-19. J Bone Joint Surg Am. 2020 Jul 15;102(14):1197-1204. doi: 10.2106/JBJS.20.00847. PMID 32675661
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] Spruit MA, Holland AE, Singh SJ, Tonia T, Wilson KC, Troosters T. COVID-19: interim guidance on rehabilitation in the hospital and post-hospital phase from a European Respiratory Society- and American Thoracic Society-coordinated international task force. Eur Respir J. 2020 Dec 3;56(6):2002197. doi: 10.1183/13993003.02197-2020. Print 2020 Dec. PMID 32817258
- [Background] Jimenez-Pavon D, Carbonell-Baeza A, Lavie CJ. Physical exercise as therapy to fight against the mental and physical consequences of COVID-19 quarantine: Special focus in older people. Prog Cardiovasc Dis. 2020 May-Jun;63(3):386-388. doi: 10.1016/j.pcad.2020.03.009. Epub 2020 Mar 24. No abstract available. PMID 32220590
- [Background] Liu K, Zhang W, Yang Y, Zhang J, Li Y, Chen Y. Respiratory rehabilitation in elderly patients with COVID-19: A randomized controlled study. Complement Ther Clin Pract. 2020 May;39:101166. doi: 10.1016/j.ctcp.2020.101166. Epub 2020 Apr 1. PMID 32379637